CLINICAL TRIAL: NCT05623449
Title: Monocentric Pilot Study of the Feasibility of Teleconsultations Hypnosis Sessions Led by a Nurse for Patients with Peripheral Chronic Neuropathic Pain - HYPTEC
Brief Title: Teleconsultations Hypnosis Sessions for Patients with Peripheral Chronic Neuropathic Pain
Acronym: HYPTEC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CHUBX 2022/34
Record Dates: First submitted 2022-10-27; First posted 2022-11-21 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Peripheral Neuropathy; Pain
Keywords: peripheral chronic neuropathic pain; hypnosis; teleconsultations; feasability
MeSH Terms: conditions — Peripheral Nervous System Diseases; Pain | interventions — Restraint, Physical; Maintenance; Data Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- combination of face-to-face and teleconsultation hypnosis consultation (Experimental): The first and the last hypnosis sessions in face-to-face, and the other 3 intermediate sessions being conducted by teleconsultation.
  Interventions: Other: Clinical examination; Other: Anxiety and Depression Scale (HAD); Procedure: pain scale; Procedure: hypnosis consultation; Procedure: Maintenance; Other: Data collection
- face-to-face hypnosis consultation (Active Comparator): 5 face-to-face hypnosis sessions
  Interventions: Other: Clinical examination; Other: Anxiety and Depression Scale (HAD); Procedure: pain scale; Procedure: hypnosis consultation; Procedure: Maintenance; Other: Data collection

INTERVENTIONS:
Other: Clinical examination — Current medications (only those prescribed to treat pain, anxiety and depression), non-drug treatment(s) prior to treatment in hypnosis as well as any ongoing treatment(s).
Other: Anxiety and Depression Scale (HAD) — To screen for anxious and depressive symptoms
Procedure: pain scale — Measurement of pain intensity
Procedure: hypnosis consultation — 5 hypnosis consultation
Procedure: Maintenance — Qualitative assessment
Other: Data collection — Age, sex, socio-professional category, level of education, comorbidities, date of diagnosis of chronic peripheral neuropathic pain, distance between home and hospital.

SUMMARY:
The aim of this study is to assess the feasibility of hypnosis sessions performed in teleconsultations and led by a nurse, for patients with peripheral chronic neuropathic pain. Acceptability, satisfaction and effects (on pain and psychological distress) are also evaluated, comparing patients who have benefited from teleconsultations and those who did not.

DETAILED DESCRIPTION:
Factors explaining peripheral chronic neuropathic pains are complex ; they require a personalized therapeutic strategy and multidisciplinary management. Among the recommended management, psychocorporal approaches such as hypnosis, are subject of recent interest. At the CHU de Bordeaux, the management of patients suffering from such chronic pains, consists of 5 hypnosis sessions, conducted face-to-face, each performed one month apart : the first session is carried out by a doctor and a hypnotherapist nurse and the 4 following sessions by the hypnotherapist nurse alone. However, it seems that this usual management is not easily accessible for patients who are geographically distant and/or who are unable to move due to excessive pain. In such situations, teleconsultations would avoid travel for these patients with low mobility and then would an interesting alternative to face-to-face consultations. Few studies have been done on hypnosis sessions led by teleconsultations. So, the whole purpose of this study is to compare the management of 15 patients by teleconsultations (experimental arm) with 15 other patients seen in face-to-face (control arm) to evaluate feasibility of teleconsultation in hypnosis.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged over 18 years old,
* Patient suffering of from peripheral neuropathic pain for more than 1 year,
* Patient referred for hypnosis management as part of a coordinated care support,
* Patient who accepts teleconsultation, having the appropriate equipment to attend teleconsultations (computer, microphone, camera and stable internet connection with sufficient internet speed) and the ability to use it independently,
* Patient having signed a free, informed and written consent,
* Patient affiliated or beneficiary of the social security system.

Exclusion Criteria:

* Patient with severe and unstable neurocognitive or psychiatric conditions (depression, psychoses, major cognitive impairments),
* Patient with uncorrected deafness,
* Patient with poor understanding of French
* Patient placed under judicial safeguard, guardianship or curatorship.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-02-23 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
5 hypnosis consultations (in face-to-face and by teleconsultation). | Month 8
  The rate (%) of included patients who have completed the 5 hypnosis consultations (in face-to-face and by teleconsultation).

SECONDARY OUTCOMES:
Achievement/Acceptability | Month 8
  Acceptance rate (%) of the proposal to participate in the study in the two study arms: face-to-face hypnosis care (control arm) and care including hypnosis teleconsultations (experimental arm).
Numerical Pain Assessme | Day 0, month 1, month 2, month 3 month 4 and montth 7
  Mean difference in pain score, minimum value is 0 and maximum value is 10
Hospital Anxiety and Depression scale (HAD) | Day 0, month 4 and month 7
  Mean difference in the anxiety and depression score, minimum value is 0 and maximum value is 42
Learning self-hypnosis | Day 0, month 1, month 2, month 3 month 4 and montth 7
  Evaluate the frequency of the use of self-hypnosis throughout the treatment.
Ssatisfaction scale | Month 7
  Evaluate the level of satisfaction and the feeling of the patients with regard to the nursing care in hypnosis at the end of the care in the two study arms (face-to-face control arm and experimental arm with teleconsultations).

CONTACTS AND LOCATIONS:
Overall Officials: Jennie SOURZAC, Principal Investigator — Université Hospital, Bordeaux
Locations (1):
- Université Hospital, Bordeaux, Pessac, Pessac, France